CLINICAL TRIAL: NCT04439318
Title: MATCH Treatment Subprotocol S1: Phase II Study of Trametinib in Patients With Tumors With NF1 Mutations
Brief Title: Testing Trametinib as a Potential Targeted Treatment in Cancers With NF1 Genetic Changes (MATCH-Subprotocol S1)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03343; NCI-2020-03343 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-S1 (Other: ECOG-ACRIN Cancer Research Group); EAY131-S1 (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib dimethyl sulfoxide PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras

SUMMARY:
This phase II MATCH treatment trial identifies the effects of trametinib in patients whose cancer has a has a genetic change called NF1 mutation. Trametinib blocks proteins called MEK1 and MEK2, which may be needed for cancer cell growth when an NF1 mutation is present. Researchers hope to learn if trametinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive trametinib dimethyl sulfoxide orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have deleterious inactivating mutations of NF-1, or another aberration, as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have NONE of the following cardiac criteria:

  * Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block).
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
* Patients must have an echocardiogram (ECHO) or a nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have a left ventricular ejection fraction (LVEF) < the institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients who previously received monoclonal antibody therapy (eg. ipilimumab, nivolumab, pembrolizumab and others) must have stopped the prior therapy for 8 or more weeks before starting on trametinib
* Patients with glioblastoma must have histologically or radiographically confirmed recurrent or progressive World Health Organization (WHO) grade 4 glioma (glioblastoma)

  * NOTE: All baseline and post-baseline disease assessments must be performed using contrast-enhanced cranial magnetic resonance spectroscopy (MRI) or contrast-enhanced computed tomography (CT) for subjects who cannot have MRI performed

Exclusion Criteria:

* Patients with a history of interstitial lung disease or pneumonitis are excluded
* Patients must not have known hypersensitivity to trametinib or compounds of similar chemical or biologic composition or to dimethyl sulfoxide (DMSO).
* Patients must not have a history or current evidence/risk of retinal vein occlusion (RVO). An eye exam is required at baseline
* Patients who previously received MEK inhibitors (including, but not limited to, trametinib, binimetinib, cobimetinib, selumetinib, RO4987655 (CH4987655), GDC-0623 and pimasertib) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-one patients were assigned to Subprotocol S1 after screening, all from screening cohort. Of the 81 patients, 50 patients were enrolled in arm S1 between March 2016 and July 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol S1, patients had to have a qualifying NF1 actionable mutation.
Groups:
- Treatment (Trametinib): Patients receive trametinib dimethyl sulfoxide 2mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Trametinib)
Started | 50
Eligible | 49
Eligible and Started Protocol Therapy (Three patients never started treatment. This is the primary analysis population.) | 46
Completed | 0
Not Completed | 50
Not completed — Ineligible | 1
Not completed — Never Started Treatment | 3
Not completed — Adverse Event | 10
Not completed — Death | 2
Not completed — Disease Progression | 25
Not completed — Other Complicating Disease | 2
Not completed — Withdrawal by Subject | 4
Not completed — Patient Refusal - Prefers Different Therapy | 1
Not completed — Non-Compliance | 1
Not completed — Still on Treatment | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 37
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for the detailed definitions of response criteria. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 46
percentage of participants | 4.3 [0.8 to 13.1]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 46
percentage of participants | 21 [12 to 34]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 46
months | 1.9 [1.8 to 3.5]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Forty-seven patients were included in the toxicity analysis (excluding three who did not receive protocol treatment).
Arm/Group | Treatment (Trametinib)
All-Cause Mortality (participants affected / at risk) | 38/50
Serious Adverse Events (participants affected / at risk) | 20/47
Other Adverse Events (participants affected / at risk) | 36/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib) (N=47)
Heart failure (Cardiac disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 5
Sudden death NOS (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Allergic reaction (Immune system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib) (N=47)
Anemia (Blood and lymphatic system disorders) | 9
Edema face (General disorders) | 3
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 15
Pain (General disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 19
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 20
Dry mouth (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 8
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 4
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT04439318/Prot_001.pdf